CLINICAL TRIAL: NCT04557397
Title: A Phase 1 Open-label 2-Part 2-Period Fixed-sequence Crossover Study To Assess The Effect Of Itraconazole, A Strong CYP3A Inhibitor, And The Effect Of Rifampin, A Strong CYP3A Inducer, On Pharmacokinetics Of Fruquintinib In Healthy Subjects
Brief Title: Fruquintinib CYP3A Inhibitor and Inducer Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hutchison Medipharma Limited (Industry)
Collaborators: Covance (Industry)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2020-013-00US2
Record Dates: First submitted 2020-09-15; First posted 2020-09-21 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2020-08

CONDITIONS: Drug Drug Interaction
Keywords: CYP3A
MeSH Terms: interventions — HMPL-013; Itraconazole; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A (Other): Subjects will receive fruquintinib, alone and with itraconazole.
  Interventions: Drug: Fruquintinib; Drug: Itraconazole
- Part B (Other): Subjects will receive fruquintinib, alone and with rifampin.
  Interventions: Drug: Fruquintinib; Drug: Rifampin

INTERVENTIONS:
Drug: Fruquintinib — oral VEGFR inhibitor
  Other Names: HMPL-013
Drug: Itraconazole — a synthetic triazole antifungal agent
  Arms: Part A
Drug: Rifampin — a semisynthetic antibiotic derivative of rifamycin SV
  Arms: Part B

SUMMARY:
A study to assess the effect of itraconazole, a strong CYP3A inhibitor, and the effect of rifampin, a strong CYP3A inducer, on the pharmacokinetics of fruquintinib in healthy subjects.

DETAILED DESCRIPTION:
This study will be a single-center, open-label, 2-part, 2-period fixed sequence crossover study to be conducted with 28 healthy male and female subjects. The study will consist of a Screening Phase (Screening and Day -1), a Treatment Phase (Period 1 and Period 2), and an End of Study (EOS) Phase. Screening will occur within 21 days before the first study drug administration. There will be at least a 14-day washout of fruquintinib between treatment periods.

Part A: subjects will be administered fruquintinib alone in treatment Period 1 and in combination with itraconazole in treatment Period 2.

Part B: subjects will be administered fruquintinib alone in treatment Period 1 and in combination with rifampin in treatment Period 2.

ELIGIBILITY:
Inclusion Criteria:

* The subject is a nonsmoking, healthy male or female between the ages of 18 and 55 years old (inclusive) at the time of informed consent.
* The subject has a body mass index (BMI) >18 and ≤29 kg/m2 at Screening.
* Females must be of non-childbearing potential (eg, postmenopausal [defined as cessation of all menstrual periods for at least 1 year confirmed by follicle-stimulating hormone (FSH) test ≥40 UI/L] or surgically sterile by total hysterectomy, bilateral oophorectomy, or bilateral tubal ligation).
* Males who have not had a successful vasectomy and are partners of women of childbearing potential must use, or their partners must use, a medically acceptable method of contraception starting for at least 1 menstrual cycle prior to and throughout the entire study period and for 2 weeks after the last dose of study drug. Those with partners using hormonal contraceptives must also use an additional approved method of contraception such as a condom with spermicide. Males who have had a successful vasectomy (confirmed azoospermia, documentation needed) require no additional contraception. No sperm donation is allowed during the study period and for 90 days after study drug discontinuation. Male subjects must confirm that female partners of childbearing potential agree to use one of the following medically accepted contraception from Screening through 2 weeks after administration of the last dose of study drug:

  1. Hormonal contraception (as the partner will not be taking the study investigational product [IP]) along with male subject's condom with spermicide
  2. Intrauterine device (hormonal or non-hormonal) along with male subject's condom with spermicide
  3. Bilateral tubal ligation
  4. Depo Provera along with male subject's condom with spermicide Abstinence is allowed (6 months of true abstinence), including same sex partners.

However, if a subject becomes sexually active during the study or, in the case of same-sex partners, has a sexual relationship with a member of the opposite sex, the subject must agree to adhere to the requirements above.

* The subject must provide written informed consent prior to any study-specific screening procedures.
* The subject is willing and able to comply with all aspects of the protocol, as determined by the investigator.

Exclusion Criteria:

* The subject has evidence of clinically significant cardiovascular, hepatic, gastrointestinal (GI), renal, respiratory, endocrine, hematological, neurological, or psychiatric diseases or abnormalities.
* The subject has a known history of any GI surgery or any condition possibly affecting drug absorption (eg, cholecystectomy, gastrectomy, achlorhydria, peptic ulcer disease, history of stomach or intestinal surgery or resection; appendectomy and hernia repair will be allowed).
* The subject had a clinically significant illness within 8 weeks or a clinically significant infection within 4 weeks prior to the first dose.
* The subject has evidence of a clinically significant deviation from normal in the physical examination, vital signs, or clinical laboratory determinations at Screening or Day -1 Check-in (baseline).
* The subject has systolic blood pressure >140 mmHg or diastolic blood pressure >90 mmHg at Screening or Day -1 Check-in (baseline).
* The subject has a clinically significant ECG abnormality, including a marked baseline prolongation of QT/QTc interval (eg, repeated demonstration of a QTcF interval >480 msec), or has a family history of prolonged QTc syndrome or sudden death.
* The subject has Gilbert's syndrome as indicated by total bilirubin > ULN and subsequent measurement of direct bilirubin is above normal range.
* The subject has a history of smoking or use of nicotine-containing substances within the previous 2 months, as determined by medical history or subject's verbal report and confirmed by cotinine test at Screening and Check-in for any one of the treatment periods.
* The subject has a history of drug or alcohol misuse within 6 months prior to Screening or a positive urine drug test at Screening or Check-in for any one of the treatment periods.
* The subject has been diagnosed with acquired immune deficiency syndrome or has performed tests that are positive for human immunodeficiency virus (HIV), Hepatitis B virus (HBV), or Hepatitis C virus (HCV).
* The subject has participated in a clinical study of other drug before screening, and the time since the last use of other study drug is less than 5 times the half-life or 4 weeks, whichever is longer, or the subject is currently enrolled in another clinical study.
* The subject has consumed grapefruit, starfruit, Seville oranges, or their products within 7 days prior to the first dose.
* The subject has consumed herbal preparations/medications, including, but not limited to kava, ephedra (ma huang), Ginkgo biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, and ginseng within 7 days prior to the first dose.
* The subject has experienced a weight loss or gain of >10% within 4 weeks prior to the first dose.
* The subject has received blood or blood products within 4 weeks, or donated blood or blood products within 8 weeks prior to the first dose or donated double red cell within 16 weeks prior to the first dose.
* The subject has used any over-the-counter (OTC) medications or prescription drugs within 2 weeks prior to the first dose.
* The subject has used CYP3A inducers (including St. John's wort) or inhibitors within 2 weeks before Day 1.
* The subject is allergic to any of the study drugs or to any of their excipients.
* The subject has used a proton pump inhibitor (PPI) within 4 days prior to the first dose or a histamine 2 (H2) receptor antagonist (H2 blocker) within 2 days prior to the first dose.
* The subject has a known allergy to azole antifungals (for Part A: itraconazole)
* The subject cannot abstain from using a PPI or an H2 blocker or locally acting antacids (eg, Gaviscon, Gelusil, Maalox, Milk of Magnesia, Mylanta, Rolaids, Tums).
* The subject has any condition that would make him or her, in the opinion of the investigator or sponsor, unsuitable for the study, or who, in the opinion of the investigator, is not likely to complete the study for any reason.
* Female subject is pregnant, lactating, or breastfeeding.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2020-10-18 (Actual); Study Completion 2020-10-18 (Actual)

PRIMARY OUTCOMES:
AUC (0-t) of fruquintinib | up to 26 days
  Pharmacokinetics of fruquintinib by assessment of area under the plasma concentration time curve from zero to the last measurable concentration
AUC (0-inf) of fruquintinib | up to 26 days
  Pharmacokinetics of fruquintinib by assessment of area under the plasma concentration curve from zero extrapolated to infinity
Cmax of fruquintinib | up to 26 days
  Pharmacokinetics of fruquintinib by assessment of maximum plasma fruquintinib concentration

SECONDARY OUTCOMES:
Number of participants with treatment emergent adverse events as assessed by CTCAE v5.0 | up to 26 days
  To evaluate the safety, in healthy subjects, of a single dose of fruquintinib administered with and without food

CONTACTS AND LOCATIONS:
Overall Officials: Youngiun Kim, MD, Principal Investigator — WCCT Global Inc
Locations (1):
- WCCT, Cypress, California, United States

IPD SHARING:
Plan to Share IPD: No